CLINICAL TRIAL: NCT04335136
Title: Recombinant Human Angiotensin-converting Enzyme 2 (rhACE2) as a Treatment for Patients With COVID-19
Acronym: APN01-COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apeiron Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APN01-01-COVID19
Record Dates: First submitted 2020-04-01; First posted 2020-04-06 (Actual); Results first posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — alunacedase alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (active) APN01 (Active Comparator): Recombinant human angiotensin-converting enzyme 2 (rhACE2) - APN01
  Interventions: Drug: RhACE2 APN01
- Group B (placebo control) (Placebo Comparator)
  Interventions: Drug: Physiological saline solution

INTERVENTIONS:
Drug: RhACE2 APN01 — Patients will be treated with APN01 intravenously twice daily (BID).
  Other Names: APN01; Recombinant human angiotensin-converting enzyme 2
  Arms: Group A (active) APN01
Drug: Physiological saline solution — Patients will be treated with placebo intravenously twice daily (BID).
  Arms: Group B (placebo control)

SUMMARY:
Recombinant human angotensin-converting enzyme 2 (rhACE2) as a treatment for patients with COVID-19 to block viral entry and decrease viral replication.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized male or female
2. Diagnosed to be COVID-19 POSITIV
3. Signed Inform Consent Form

Exclusion Criteria:

1. Any patient whose clinical condition is deteriorating rapidly
2. Known history of positive Hepatitis B surface antigen, Hepatitis C antibody or HIV antibody
3. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation
4. Pregnant females as determined by positive serum or urine hCG test prior to dosing
5. Lung transplantation
6. Pre-existing renal failure, i.e. requiring renal replacement therapy with hemodialysis or peritoneal dialysis
7. There are other uncontrolled co-morbidities that increase the risks associated with the study drug administration, that are assessed by the medical expert team as unsuitable
8. Patient in clinical trials for COVID-19 within 30 days before ICF
9. Immunocompromised patients (chemotherapy, HIV, organ transplants, stem cell transplants)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-12-26 (Actual); Study Completion 2020-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henning Bundgaard, MD., Principal Investigator — Cap. Region's Unit of Inherited Cardiac Diseases, Faculty Health&Medical
Locations (22):
- Austria (3):
  - Medizinische Universität Innsbruck, Innsbruck
  - Kaiser Franz Josef Spital, 4. Medizinische Abteilung mit Infektions- und Tropenmedizin, Vienna
  - Medizinische Universität Wien, Vienna
- Denmark (4):
  - The National University Hospital, Rigshospitalet, Copenhagen
  - Herlev Gentofte Hospital, Herlev
  - Nordsjællands Hospital, Hillerød
  - Hvidovre Hospital, Hvidovre
- Germany (2):
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Klinikum rechts der Isar, Technische Universität München, München
- Russia (12):
  - Regional State Budgetary Educational Institution "Clinical Hospital № 5, Barnaul", Barnaul
  - State Healthcare Institution "State Clinical Hspital № 15 named after O.M. Filatov", Moscow
  - Moscow State Budgetary Healthcare Institution "City Clinical Hospital №52 of Health Department of Moscow", Moscow
  - Moscow State Budgetary Healthcare Institution "N.V. Sklifosovsky Research Institute for Emergency Medicine of Health Department of Moscow", Moscow
  - Saint Petersburg SBHI City Hospital 38 named after N A Semashko, Pushkin
  - Federal State Budgetary Educational Institution of Higher Education "Ryazan State Medical University named after I.P. Pavlov" HD RF, Ryazan
  - Alexandrovskaya Hospital, Saint Petersburg
  - Saint-Petersburg State Budget Healthcare Institution City Hospital 15, Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education " Saratov State Medical University named after V.I. Razumovsky" HD RF, Saratov
  - Regional State Budgetary Healthcare Institution "Clinical Hospital №1", Smolensk
  - State budgetary institution of Healthcare of Tver region "Regional clinical hospital", Tver'
  - Yaroslavl Regional Clinical Hospital for Military Veterans - International Centre for Gerontological Problems "Healthy Ageing", Yaroslavl
- Cambridge University Hospitals NHS Trust/University of Cambridge, Cambridge, United Kingdom

REFERENCES:
- [Derived] Chene A, Desrames A, Tomlinson A, Ruffie C, Tangy F, Gamain B. An ACE2-Based Bimodular Fusion Protein Enables Reorientation of Endogenous Anti-Epstein-Barr Virus Antibodies Toward SARS-CoV-2 Spike. J Infect Dis. 2023 Dec 20;228(12):1675-1679. doi: 10.1093/infdis/jiad329. PMID 37562051
- [Derived] Morrell ED. Tipping the Balance of Ubiquitination toward a Therapy for COVID-19. Am J Respir Cell Mol Biol. 2023 May;68(5):480-481. doi: 10.1165/rcmb.2023-0020ED. No abstract available. PMID 36796097

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 185 Patients were screened of whom 181 patients were randomized.
Groups:
- Group A (Active) APN01: Patients were treated with APN01 (Recombinant human angiotensin-converting enzyme 2 [rhACE2]) intravenously twice daily (BID).
- Group B (Placebo Control): Patients were treated with placebo (physiological saline solution) intravenously twice daily (BID).
Period: Overall Study
Arm/Group | Group A (Active) APN01 | Group B (Placebo Control)
Started (Patients randomized.) | 91 | 90
Treated | 88 | 90
Completed | 77 | 83
Not Completed | 14 | 7
Not completed — Death | 8 | 4
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Health-threatening condition | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Erroneously randomized | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients who received at least 1 dose of investigational medicinal product (IMP).
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Active) APN01 | Group B (Placebo Control) | Total
Number analyzed (Participants) | 88 | 90 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (11.3) | 58.5 (12.4) | 59.0 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 64
  Male | 55 | 59 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 88 | 90 | 178
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data of 1 patient in the placebo group are missing.
  Participants
    number analyzed (Participants) | 88 | 89 | 177
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 0 | 1
    White | 86 | 88 | 174
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 19 | 20 | 39
  Germany | 2 | 3 | 5
  Russia | 67 | 67 | 134

OUTCOME MEASURES:

1. Primary Outcome: All Cause-death or Invasive Mechanical Ventilation
Description: The primary endpoint was a composite endpoint of all cause-death or invasive mechanical ventilation up to 28 days or hospital discharge.
Time Frame: 28 days
Population: All randomized patients who had received at least 1 dose of investigational medicinal product (IMP).
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Active) APN01 | Group B (Placebo Control)
Number analyzed (Participants) | 88 | 90
Participants | 9 | 12
Statistical Analysis 1: Comparison: Group A (Active) APN01 vs Group B (Placebo Control); Hypothesis tested: H0: pAPN01 = pPlacebo; H1: pAPN01 ≠ pPlacebo (with p=proportion of patients with event). A total of 186 patients (93 per group) was estimated to yield 80% power to detect a 20% absolute risk reduction in the primary, from 50% in the placebo group to 30% in the APN01 group, at a 2-sided alpha of 0.05. To consider patients who would be randomized but not treated, a total of 200 patients (100 per group) were planned to be enrolled; Test type: Other; p = 0.5207, Chi-squared — The level of significance was 5% (2-sided)
Statistical Analysis 2: Comparison: Group A (Active) APN01 vs Group B (Placebo Control); Test type: Other; p = 0.3588, Regression, Logistic; Degree of freedom: 1; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.23 to 1.70]

2. Secondary Outcome: Lactate Dehydrogenase (LDH) Level
Description: Log transformed levels of LDH at Day 5 as a surrogate marker for organ damage (powered secondary endpoint).
Time Frame: Day 5
Population: All randomized patients who had received at least 1 dose of IMP and had an LDH measurement at Day 5.
Measure: Mean (Standard Deviation); unit: Log U/L
Arm/Group | Group A (Active) APN01 | Group B (Placebo Control)
Number analyzed (Participants) | 74 | 74
Log U/L | 5.82 (0.470) | 5.80 (0.433)

3. Secondary Outcome: Mortality
Description: 28-day mortality (all cause-death).
Time Frame: 28 days
Population: All randomized patients who had received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Active) APN01 | Group B (Placebo Control)
Number analyzed (Participants) | 88 | 90
Participants | 9 | 7

4. Secondary Outcome: Ventilator-free Days (VFD)
Description: VFD up to 28 days or hospital discharge. VFD and mechanical-VFD (mVFD) were calculated as time in the study minus duration of ventilation and were set to zero if the duration of ventilation exceeded the time in the study.
  Three analysis approaches were used: 1) Death not censored: (m)VFD was set to zero for patients who died. 2) Death censored: patients who died before or on Day 28 were censored at the day before death. 3) Alive patients analyzed: only patients who were alive at Day 28, hospital discharge, or early termination were included in the analysis.
Time Frame: 28 days
Population: All randomized patients who had received at least 1 dose of IMP. In addition, a subgroup analysis was performed including only patients who were still alive at Day 28 (or discharged from the hospital/early terminated).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group A (Active) APN01 | Group B (Placebo Control)
Number analyzed (Participants) | 88 | 90
days
  VFD (death not censored) | 17.2 (8.8) | 16.7 (8.4)
  VFD (death censored) | 17.4 (8.6) | 16.7 (8.4)
  VFD (subgroup: alive patients): number analyzed (Participants) | 80 | 84
  VFD (subgroup: alive patients) | 18.9 (7.3) | 17.9 (7.4)
  mVFD (death not censored) | 25.7 (8.4) | 25.1 (8.7)
  mVFD (death censored) | 26.3 (6.6) | 25.6 (7.6)
  mVFD (subgroup: alive patients): number analyzed (Participants) | 79 | 83
  mVFD (subgroup: alive patients) | 28.2 (1.9) | 26.9 (5.8)

5. Secondary Outcome: Time to Death
Description: Time to death (all causes).
Time Frame: 28 days
Population: All randomized patients who had received at least 1 dose of IMP.
Measure: Median (Full Range); unit: days
Arm/Group | Group A (Active) APN01 | Group B (Placebo Control)
Number analyzed (Participants) | 88 | 90
days | NA [6 to 22] — Median time to death could not be estimated due to an insufficient number of patients with events. | NA [2 to 28] — Median time to death could not be estimated due to an insufficient number of patients with events.

6. Secondary Outcome: Number of Responders, Defined as ≥2 Improvement in World Health Organization (WHO)'s 11-Point Score System at Days 7, 10, 14 and 28
Description: The WHO Clinical Progression Scale provides a measure of illness severity across an 11 point range from 0 (not infected) to 10 (dead) as follows (scores 4-9 contain measures of respiratory failure):
  Uninfected, no viral deoxyribonucleic acid (DNA) detected = 0;
  Asymptomatic, viral DNA detected = 1;
  Symptomatic, independent = 2;
  Symptomatic, assistance needed = 3;
  Hospitalized, no oxygen therapy = 4;
  Hospitalized, oxygen by mask or nasal prongs = 5;
  Hospitalized, oxygen by non-invasive ventilation (NIV) or high flow = 6;
  Intubation and mechanical ventilation, partial pressure of oxygen (pO2)/fraction of inspired oxygen (FiO2)≥ 150 or oxygen saturation (SpO2)/FiO2≥200 = 7;
  Mechanical ventilation, pO2/FiO2 < 150 (SpO2/FiO2 < 200) or vasopressors = 8;
  Mechanical ventilation, pO2/FiO2 < 150 and vasopressors, dialysis, or extracorporeal membrane oxygenation (ECMO) = 9;
  Dead = 10.
  A decrease in the score reflects an improvement.
Time Frame: Day 7, Day 10, Day 14, Day 28
Population: All randomized patients who had received at least 1 dose of IMP and who had a measurement of the WHO 11-Point Score System at the respective timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Active) APN01 | Group B (Placebo Control)
Number analyzed (Participants) | 88 | 90
Participants
  Day 7: number analyzed (Participants) | 88 | 88
  Day 7 | 2 | 0
  Day 10: number analyzed (Participants) | 86 | 85
  Day 10 | 17 | 13
  Day 14: number analyzed (Participants) | 83 | 85
  Day 14 | 38 | 32
  Day 28: number analyzed (Participants) | 79 | 83
  Day 28 | 72 | 74

7. Secondary Outcome: Time to Hospital Discharge
Description: The number of days from randomization to discharge from hospital was calculated (Kaplan-Meier analysis).
  Patients without hospitalization or without documented hospital discharge who completed the study or were early terminated before Day 28 were censored at the date of study completion or discontinuation, respectively.
  Patients who died before Day 28 were censored at the date of death even if early terminated before.
Time Frame: Up to 28 days
Population: All patients who had received at least 1 dose of IMP.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Group A (Active) APN01 | Group B (Placebo Control)
Number analyzed (Participants) | 88 | 90
days | 14 [12 to 15] | 14 [13 to 15]

8. Secondary Outcome: Viral Ribonucleic Acid (RNA).
Description: Viral RNA was assessed in blood samples using quantitative reverse transcriptase polymerase chain reaction (RT-PCR) and projected to RNA copies per mL.
Time Frame: Day 1, Day 3, Day 5, Day 7, Day 14, and Day 28/End of study (EOS)
Population: All randomized patients who had received at least 1 dose of IMP and who had a measurement of viral RNA at the respective timepoint.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Group A (Active) APN01 | Group B (Placebo Control)
Number analyzed (Participants) | 88 | 90
copies/mL
  Day 1: number analyzed (Participants) | 59 | 49
  Day 1 | 27996 (78877) | 3900 (5848)
  Day 3: number analyzed (Participants) | 47 | 58
  Day 3 | 20931 (53182) | 13681 (45287)
  Day 5: number analyzed (Participants) | 56 | 64
  Day 5 | 9825 (32979) | 11912 (75457)
  Day 7: number analyzed (Participants) | 65 | 61
  Day 7 | 5229 (24514) | 2094 (8742)
  Day 14: number analyzed (Participants) | 73 | 73
  Day 14 | 9274 (78304) | 53 (455)
  Day 28/EOS: number analyzed (Participants) | 37 | 0
  Day 28/EOS | 36 (217) |

9. Secondary Outcome: Time to a 2-point Decrease in WHO's 11-Point Score System
Description: The time from randomization to an at least 2-point decrease in the WHO scale was calculated. The WHO Clinical Progression Scale provides a measure of illness severity across an 11 point range from 0 (not infected) to 10 (dead) as follows (scores 4-9 contain measures of respiratory failure):
  Uninfected, no viral DNA detected = 0;
  Asymptomatic, viral DNA detected = 1;
  Symptomatic, independent = 2;
  Symptomatic, assistance needed = 3;
  Hospitalized, no oxygen therapy = 4;
  Hospitalized, oxygen by mask or nasal prongs = 5;
  Hospitalized, oxygen by non-invasive ventilation (NIV) or high flow = 6;
  Intubation and mechanical ventilation, pO2/FiO2 ≥ 150 or SpO2/FiO2≥200 = 7;
  Mechanical ventilation, pO2/FiO2 < 150 (SpO2/FiO2 < 200) or vasopressors = 8;
  Mechanical ventilation, pO2/FiO2 < 150 and vasopressors, dialysis, or ECMO = 9;
  Dead = 10.
  A decrease in the score reflects an improvement in disease status.
Time Frame: Up to 28 days.
Population: All randomized patients who had received at least 1 dose of IMP.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Group A (Active) APN01 | Group B (Placebo Control)
Number analyzed (Participants) | 88 | 90
days | 27 [14 to 27] | 27 [17 to 27]

10. Secondary Outcome: Number of Patients With Any Use of Invasive Mechanical Ventilation up to 28 Days or Hospital Discharge
Description: The number of patients receiving mechanical ventilation and supplemental oxygen was evaluated.
Time Frame: Up to 28 days
Population: All randomized patients who had received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Active) APN01 | Group B (Placebo Control)
Number analyzed (Participants) | 88 | 90
Participants
  Mechanical ventilation | 7 | 7
  Mechanical ventilation and oxygen supplementation | 86 | 88

11. Secondary Outcome: Time to First Use of Invasive Mechanical Ventilation up to 28 Days or Hospital Discharge
Description: Time from randomization to first use of invasive mechanical ventilation was calculated (Kaplan-Meier analysis).
  Patients without documented invasive mechanical ventilation who completed the study, were early terminated or discharged from hospital before Day 28 were censored at the date of study completion, discontinuation or discharge from hospital, respectively.
Time Frame: Up to 28 days
Population: All randomized patients who had received at least 1 dose of IMP.
Measure: Median (Full Range); unit: days
Arm/Group | Group A (Active) APN01 | Group B (Placebo Control)
Number analyzed (Participants) | 88 | 90
days | NA [0 to 14] — Median time to first invasive mechanical ventilation could not be estimated due to an insufficient number of patients with events. | NA [0 to 20] — Median time to first invasive mechanical ventilation could not be estimated due to an insufficient number of patients with events.

12. Secondary Outcome: PaO2/FiO2 Value
Description: The ratio in partial pressure of arterial oxygen (PaO2)/fraction of inspired oxygen (FiO2) was assessed by analysis of patient's blood gas.
Time Frame: Day 1, Day 7, Day 10, Day 14, and Day 28
Population: All randomized patients who had received at least 1 dose of IMP and who had a measurement of PaO2/FiO2 at the respective timepoint.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group A (Active) APN01 | Group B (Placebo Control)
Number analyzed (Participants) | 88 | 90
mmHg
  Day 1: number analyzed (Participants) | 30 | 28
  Day 1 | 223.07 (99.70) | 185.14 (79.79)
  Day 7: number analyzed (Participants) | 19 | 24
  Day 7 | 218.74 (91.66) | 192.21 (92.71)
  Day 10: number analyzed (Participants) | 14 | 13
  Day 10 | 290.00 (204.70) | 186.62 (87.83)
  Day 14: number analyzed (Participants) | 9 | 11
  Day 14 | 197.00 (99.42) | 185.00 (67.20)
  Day 28: number analyzed (Participants) | 1 | 3
  Day 28 | 261.00 (NA) — Data of only 1 patient were available. | 185.00 (116.73)

13. Secondary Outcome: Modified Sequential Organ Failure Assessment Score (mSOFA Score, Total Score)
Description: The mSOFA score predicts intensive care unit mortality using clinical and laboratory variables. 5 organ systems (respiratory SpO2/FiO2; liver; cardiovascular/hypotension; Central nervous System/Glasgow Coma Score; renal/creatinine), all, except for liver, scored on a 0 to 4 scale (liver: 2-point scale: 0 or 3) according to specified criteria indicating severity, with the total score ranging from 0 to a maximum score of 19. A higher score reflects a worse disease state.
Time Frame: Day -1 (Screening), Day 7, Day 10, Day 14, Day 28/End of study
Population: All randomized patients who had received at least 1 dose of IMP and who had a measurement of the mSOFA score at the respective timepoint.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Group A (Active) APN01 | Group B (Placebo Control)
Number analyzed (Participants) | 88 | 90
score on a scale
  Day -1: number analyzed (Participants) | 80 | 80
  Day -1 | 2.6 (1.2) | 2.2 (1.4)
  Day 7: number analyzed (Participants) | 83 | 77
  Day 7 | 1.8 (2.5) | 1.6 (2.1)
  Day 10: number analyzed (Participants) | 80 | 77
  Day 10 | 1.0 (1.7) | 1.0 (1.6)
  Day 14: number analyzed (Participants) | 79 | 75
  Day 14 | 1.0 (2.4) | 0.9 (1.7)
  Day 28/EOS: number analyzed (Participants) | 39 | 38
  Day 28/EOS | 0.2 (0.6) | 0.8 (1.8)

14. Secondary Outcome: Lymphocyte Count
Description: Lymphocytes were assessed in blood samples from the patients.
Time Frame: Day -1, Day 3, Day 7, Day 10, Day 14, Day 28/End of study
Population: All randomized patients who had received at least 1 dose of IMP and who had a measurement of lymphocyte count at the respective timepoint.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Group A (Active) APN01 | Group B (Placebo Control)
Number analyzed (Participants) | 88 | 90
10^9 cells/L
  Day -1: number analyzed (Participants) | 82 | 82
  Day -1 | 1.13 (0.694) | 1.06 (0.629)
  Day 3: number analyzed (Participants) | 85 | 83
  Day 3 | 1.25 (0.843) | 1.16 (0.662)
  Day 7: number analyzed (Participants) | 82 | 80
  Day 7 | 1.45 (0.948) | 1.62 (0.940)
  Day 10: number analyzed (Participants) | 81 | 75
  Day 10 | 1.74 (1.444) | 1.79 (0.782)
  Day 14: number analyzed (Participants) | 77 | 73
  Day 14 | 1.70 (0.773) | 1.71 (0.730)
  Day 28/EOS: number analyzed (Participants) | 37 | 37
  Day 28/EOS | 2.28 (3.420) | 1.72 (0.559)

15. Secondary Outcome: C-reactive Protein Levels
Description: C-reactive protein was assessed in blood samples from the patients.
Time Frame: Day -1, Day 3, Day 7, Day 10, Day 14, Day 28/End of study
Population: All randomized patients who had received at least 1 dose of IMP and who had a C-reactive protein measurement at the respective timepoint.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Group A (Active) APN01 | Group B (Placebo Control)
Number analyzed (Participants) | 88 | 90
mg/L
  Day -1: number analyzed (Participants) | 77 | 79
  Day -1 | 56.0 (64.53) | 62.8 (51.75)
  Day 3: number analyzed (Participants) | 80 | 74
  Day 3 | 36.1 (53.75) | 43.7 (45.13)
  Day 7: number analyzed (Participants) | 78 | 76
  Day 7 | 21.7 (41.58) | 26.1 (38.71)
  Day 10: number analyzed (Participants) | 74 | 71
  Day 10 | 13.9 (24.24) | 26.3 (48.75)
  Day 14: number analyzed (Participants) | 69 | 73
  Day 14 | 15.8 (29.66) | 38.3 (133.24)
  Day 28/EOS: number analyzed (Participants) | 36 | 37
  Day 28/EOS | 4.9 (5.69) | 8.5 (11.54)

16. Secondary Outcome: D-Dimer
Description: D-Dimer was assessed in blood samples from the patients.
Time Frame: Day -1, Day 3, Day 7, Day 10, Day 14, Day 28/End of study
Population: All randomized patients who had received at least 1 dose of IMP and who had a D-Dimer measurement at the respective timepoint.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Group A (Active) APN01 | Group B (Placebo Control)
Number analyzed (Participants) | 88 | 90
µg/L
  Day -1: number analyzed (Participants) | 71 | 73
  Day -1 | 1341 (2757) | 1187 (3994)
  Day 3: number analyzed (Participants) | 69 | 74
  Day 3 | 1109 (1316) | 881 (959)
  Day 7: number analyzed (Participants) | 73 | 68
  Day 7 | 1208 (1485) | 1139 (1590)
  Day 10: number analyzed (Participants) | 70 | 66
  Day 10 | 988 (1135) | 1219 (2228)
  Day 14: number analyzed (Participants) | 70 | 66
  Day 14 | 1015 (1520) | 1013 (2243)
  Day 28/EOS: number analyzed (Participants) | 32 | 31
  Day 28/EOS | 573 (629) | 685 (939)

17. Secondary Outcome: Log-transformed Levels of LDH
Description: Log transformed levels of LDH in blood were assessed as a surrogate marker for organ damage.
Time Frame: Day -1, Day 3, Day 7, Day 10, Day 14, Day 28/End of study
Population: All randomized patients who had received at least 1 dose of IMP and who had an LDH measurement at the respective timepoints.
Measure: Mean (Standard Error); unit: Log U/L
Arm/Group | Group A (Active) APN01 | Group B (Placebo Control)
Number analyzed (Participants) | 88 | 90
Log U/L
  Day -1: number analyzed (Participants) | 78 | 77
  Day -1 | 5.91 (0.442) | 5.87 (0.489)
  Day 3: number analyzed (Participants) | 76 | 76
  Day 3 | 5.86 (0.440) | 5.88 (0.422)
  Day 7: number analyzed (Participants) | 78 | 74
  Day 7 | 5.77 (0.459) | 5.75 (0.387)
  Day 10: number analyzed (Participants) | 72 | 74
  Day 10 | 5.66 (0.464) | 5.67 (0.401)
  Day 14: number analyzed (Participants) | 69 | 71
  Day 14 | 5.55 (0.467) | 5.52 (0.406)
  Day 28/EOS: number analyzed (Participants) | 38 | 38
  Day 28/EOS | 5.43 (0.305) | 5.50 (0.383)

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Group A (Active) APN01 | Group B (Placebo Control)
All-Cause Mortality (participants affected / at risk) | 9/88 | 7/90
Serious Adverse Events (participants affected / at risk) | 10/88 | 12/90
Other Adverse Events (participants affected / at risk) | 14/88 | 24/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Active) APN01 (N=88) | Group B (Placebo Control) (N=90)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7)
Infarction (Vascular disorders) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Active) APN01 (N=88) | Group B (Placebo Control) (N=90)
Alanine aminotransferase increased (Investigations) | 10 (10) | 11 (11)
Blood potassium increased (Investigations) | 5 (5) | 4 (4)
Electrocardiogram QT prolonged (Investigations) | 2 (2) | 6 (6)
Hepatic enzyme increased (Investigations) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT04335136/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/36/NCT04335136/SAP_001.pdf